CLINICAL TRIAL: NCT05284773
Title: Screening for Acute Malnutrition: a Cluster Randomized Trial Comparing Caregivers to Community Health Workers in Burkina Faso
Brief Title: Screening for Acute Malnutrition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding for recruitment of participants
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-24230
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Malnutrition in Childhood

STUDY DESIGN:
Intervention Model Description: One group will be randomized to intervention + standard of care; one group will be randomized to standard of care only
Who Masked: Outcomes Assessor
Masking Description: Masking of participants and intervention administrators will not be possible due to the nature of the intervention. Primary outcome assessors will be masked to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention + standard of care (Experimental): Caretakers of children 6-59 months old living in communities assigned to the intervention arm will be trained to detect malnutrition using MUAC on their children weekly. Caretakers living in communities assigned to the intervention will also receive usual standard of care.
  Interventions: Other: Caretaker MUAC screening - training by health workers; Other: Caretaker MUAC screening - training by caregivers
- standard of care (No Intervention): Caretakers of children 6-59 months living in communities assigned to the standard of care arm will receive usual acute malnutrition screening. This includes biannual community-based screening by community health workers as well as weekly malnutrition days led by the Centre de Sante et Promotion Sociale (CSPS).

INTERVENTIONS:
Other: Caretaker MUAC screening - training by health workers — Study personnel will train caregivers to conduct weekly AM screening using the color-coded MUAC tape. AM screening will involve identifying the midpoint of the child's right arm, wrapping the tape around the mid-point, inserting one end of the tape through the slit at the other end, pulling the tape secure, and reading the measurement based on the color bands. Caregivers will be trained to refer children with yellow or red readings to the nearest CSPS and will be provided with a referral slip to do so. Caregivers will be informed of the signs, symptoms, and consequences of malnutrition as well as the available nutritional programs. Study personnel will conduct monthly supervision visits including brief refresher trainings. In all study communities, standard of care screening for AM will continue. This includes biannual community-based screening by community health workers as well as weekly malnutrition days led by the CSPS.
  Arms: intervention + standard of care
Other: Caretaker MUAC screening - training by caregivers — Study personnel will train a group of caregivers to perform AM training of all caregivers living in their communities. they will instruct caregivers to conduct weekly AM screening. Training will include the same information as the communities receiving training by Health workers: MUAC training and how to interpret MUAC as well as key concepts of malnutrition. Caregivers will be trained to refer children with yellow or red readings to the nearest CSPS and will be. In all study communities, standard of care screening for AM will continue. This includes biannual community-based screening by community health workers as well as weekly malnutrition days led by the CSPS.
  Arms: intervention + standard of care

SUMMARY:
This project includes a pilot cluster-randomized trial of the efficacy of training caregivers to screen for acute malnutrition (AM) in children aged 6-59 months using mid-upper arm circumference (MUAC) in Burkina Faso. The pilot will be conducted to establish the feasibility of procedures and preliminary outcome data to inform the sample size calculations and design of a future longer-term, fully powered cluster-randomized trial. Forty communities enrolled in the Bill & Melinda Gates Foundation-funded Child Health with Azithromycin Treatment (CHAT) trial will be randomly selected for this pilot and randomized to receive the caregiver training intervention or no additional intervention. All communities will continue to receive standard of care screening for AM according to national guidelines, which includes community-based screening for AM by community health workers using MUAC every 6 months. A baseline census will be conducted before randomization to enumerate the eligible population of caregivers and children 6-59 months old and measure MUAC. A final census with MUAC measurement will be conducted 6 months later (primary outcome). Data will be collected on all children presenting to the Centre de Santé et Promotion Sociale (CSPS) for malnutrition to track secondary outcomes.

During intervention training, we will also conduct a diagnostic accuracy study to evaluate the validity of caregiver screening by comparing the MUAC measurements of caregivers against the gold standard measurement of the experienced health personnel conducting the training. Also during training, intervention communities will be randomized to one of two training approaches: training by caregivers or training by health agents and adherence to the protocol during follow-up monitoring visits will be compared to determine effectiveness of training.

ELIGIBILITY:
Cluster level:

* Enrollment in the CHAT trial
* Location outside of the Health and Demographic Surveillance System (HDSS)
* Population size < 2000 people
* Verbal consent of the village leader

Individual level:

* Residence in a village participating in the CHAT trial
* Caregiver or guardian of children aged 6-59 months (for intervention training)
* Age 6-59 months (for MUAC screening and some outcome assessments)
* Verbal consent from caregiver or guardian

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2030-02-15 (Estimated); Primary Completion 2035-03-10 (Estimated); Study Completion 2035-03-10 (Estimated)

PRIMARY OUTCOMES:
Community-level mean mid-upper arm circumference (MUAC) | 6 months
  Community-level mean MUAC in children 6-59 months of age as assessed during the final census after 6 months of intervention

SECONDARY OUTCOMES:
Sensitivity | 6 months
  Diagnostic accuracy study comparing caregiver measurements to the gold standard measurement from study personnel will include sensitivity as an outcome measure, defined as the number of true positives divided by the total number of cases of global acute malnutrition (MUAC < 125 mm)
Specificity | 6 months
  Diagnostic accuracy study comparing caregiver measurements to the gold standard measurement from study personnel will include specificity as an outcome measure, defined as the number of true negatives divided by the total number of children without global acute malnutrition (MUAC < 125 mm)
Cases referred | 6 months
  Number of cases of AM referred to the CSPS during the study period as collected at the CSPS
Mid-upper arm circumference (MUAC) at admission | 6 months
  MUAC among children 6-59 months of age at admission to CSPS nutritional programs during the study period as routinely collected at the CSPS
Effectiveness of caregiver training | 6 months
  Adherence to protocol in the communities with caretakers training compared to health workers training as measured by caregiver survey and supervisor monitoring checklist. Relevant items from each data collection source will be summarized into a single summary score.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenbrug, ScD, Principal Investigator — University of California, San Francisco; Kieran O'Brien, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No